CLINICAL TRIAL: NCT00938691
Title: Optimal Suture Choice for Improved Scar Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Ponciano Cruz, MD, Chair, Division of Dermatology
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ASDS-45322
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Cicatrix
Keywords: Scar; Appearance; Spread
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tepha (Experimental)
  Interventions: Procedure: Intradermal Suture
- Vicryl (Active Comparator)
  Interventions: Procedure: Intradermal Suture

INTERVENTIONS:
Procedure: Intradermal Suture
  Arms: Tepha
Procedure: Intradermal Suture
  Arms: Vicryl

SUMMARY:
Certain parts of the body, such as the chest, back, and shoulders, are notorious for producing cosmetically poor scars after cutaneous surgery. While very little research has been done to understand these poor outcomes, it is generally thought that increased tension across the skin inherent to these body areas leads to significant widening of the final scar. Historically, the only way to combat this tension was to support the deeper portion of the wound with sutures that dissolve over several weeks. However, scars take many months to fully develop their greatest strength. So even with the standard technique, wounds in areas of high tension still show spreading of the scar with time. The investigators believe that these wounds require an extended duration of support throughout the scar's maturation period. Until recently, there did not exist a suture that could provide this long duration of support without also carrying the risk of the body rejecting it. Recently, a new extremely long acting absorbable biomaterial has been FDA approved for use as a suture. The investigators plan to use this suture to test the theory that alleviating stress on high tension wounds throughout the period which they gain their maximal integrity produces less scar spread and ultimately better cosmetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring excision of a lesion on chest, back, or shoulders

Exclusion Criteria:

* History of ionizing radiation
* History of keloid or hypertrophic scarring
* History of or current internal malignancy
* History of bleeding disorder
* History of collagen or elastin disorder
* Current use of immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Scar spread | 3 months and 1 year

SECONDARY OUTCOMES:
Scar appearance | 3 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Kia, MD, Study Director — Dermatology, UT-Southwestern
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Kia KF, Burns MV, Vandergriff T, Weitzul S. Prevention of scar spread on trunk excisions: a rater-blinded randomized controlled trial. JAMA Dermatol. 2013 Jun;149(6):687-91. doi: 10.1001/jamadermatol.2013.3004. PMID 23752288